CLINICAL TRIAL: NCT05991180
Title: Real-World Study on the Efficacy of IBI-322 in Combination With Lenvatinib for the Treatment of Extensive Stage Small Cell Lung Cancer and Assessment of Biomarkers
Brief Title: Real-World Study on the Efficacy of IBI-322 in Combination With Lenvatinib for the Treatment of Extensive Stage Small Cell Lung Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hunan Province Tumor Hospital (Other)
Responsible Party: Principal Investigator, Yongchang Zhang, Professor, Deputy Director of Thoracic Oncology Department, Hunan Province Tumor Hospital
Other Study IDs: BELIEVE RWS
Record Dates: First submitted 2023-08-06; First posted 2023-08-14 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Extensive-stage Small-cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — needle biopsy for samples with DNA
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a descriptive observational study, in which data are collected in an epidemiological fashion and prospective. This study does not intend to intervene the current medical practice of the recruited patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be ≥18 years.
* Provision of fully informed consent prior to any study specific procedures.
* Patients with extensive stage SCLC diagnosed by pathology (as staged by the American Veterans Lung Cancer Association (VALG)), who do not have an imaging response during first-line treatment with PD-(L)1 inhibitors, or who progress after imaging reactions on first-line therapy (the most recent regimen prior to enrollment must contain PD-(L)1 inhibitors).
* According to the RECIST 1.1 standard, the patient must have at least one measurable lesion.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Extensive Stage Small Cell Lung Cancer
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2023-12-25 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
ORR | 2 years
  Defined as the proportion of subjects in complete remission (CR) and partial remission (PR) to the total subjects

SECONDARY OUTCOMES:
PFS | 2 years
  Defined as the time from the beginning of treatment to the first imaging disease progression or death (whichever occurs first)
OS | 2 years
  Defined as the time from the start of treatment to the death of the subject due to any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan Cancer hospital, Changsha, Hunan, China